CLINICAL TRIAL: NCT06464679
Title: An Exploratory Clinical Study of the Safety and Efficacy of CD19 Chimeric Antigen Receptor NK Cell Injection for the Treatment of Relapsed/Refractory Autoimmune Diseases
Brief Title: An Exploratory Clinical Study of CD19 CAR NK Cell Injection for the Treatment of Relapsed/Refractory Autoimmune Diseases
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Changhai Hospital (Other)
Collaborators: Rui Therapeutics (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHEC2024-181
Record Dates: First submitted 2024-06-13; First posted 2024-06-18 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-06

CONDITIONS: Autoimmune Diseases
MeSH Terms: conditions — Autoimmune Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD19 CAR NK cells (Experimental)
  Interventions: Biological: anti-CD19 CAR NK cells

INTERVENTIONS:
Biological: anti-CD19 CAR NK cells — Patients will receive Fludarabine (25 mg/m2 per day) and Cyclophosphamide (300mg/m2 per day) on day -5, -4, and -3. Multiple doses of CD19 CAR NK cells will infused using the dose-escalation strategy.

SUMMARY:
A single arm, open-label pilot study is designed to determine the safety and effectiveness of CD19 CAR NK cells in patients with autoimmune diseases. 36-72 patients are planned to be enrolled in the dose-escalation trial. The primary objective of the study was to evaluate the safety and feasibility of CD19 CAR-NK cells for the treatment of patients with autoimmune diseases. The secondary objective is to evaluate the efficacy of CD19 CAR-NK cells in patients with autoimmune diseases.

ELIGIBILITY:
Common inclusion criteria:

1. Age: ≥ 18 years old and ≤ 65 years old, male or female;
2. The functions of important organs meet the following requirements:

<!-- -->

1. Bone marrow hematopoietic function needs to meet: a. White blood cell count ≥ 3 x 10^9/L b. Neutrophil count ≥ 1 x 10^9/L (no colony-stimulating factor treatment within 2 weeks before examination); c. Hemoglobin ≥60g/L;
2. Liver function:ALT ≤ 3 x ULN,AST≤3 x ULN, TBIL≤1.5 x ULN(excluding Gilbert syndrome, total bilirubin ≤ 3.0 x ULN) (No requirements for conditions caused by the disease itself);
3. Renal function: creatinine clearance rate (CrCl) ≥ 60 ml/minute(Cockcroft/Fault formula);
4. Coagulation function: International standardized ratio (INR) < 1.5 x ULN,prothrombin time(PT) < 1.5 x ULN;
5. Cardiac function: Good hemodynamic stability. 3. Female subjects of childbearing potential and male subjects whose partner is a female of childbearing potential are required to use medically approved contraception or abstain from sex for at least 6 months during and at least 6 months after the end of the study treatment period; female subjects of childbearing potential have had a negative serum HCG test within 7 days prior to study enrollment and are not lactating; 4. Voluntarily participate in this clinical study, sign an informed consent form, have good compliance, and cooperate with follow-up.

Inclusion Criteria for Relapsing refractory dry syndrome:

1. Meets 2002 AECG criteria or 2016 ACR/EULAR classification criteria for primary dry syndrome (pSS);
2. Definition of disease activity: investigator-assessed disease ESSDAI score of 5 or higher;
3. Definition of relapsed and refractory disease: ineffective conventional treatment or relapse of disease activity after remission. Definition of routine treatment: Use of glucocorticoids (above 1mg/Kg/d) and cyclophosphamide, as well as any of the following immunomodulatory drugs for more than 6 months: antimalarials, methotrexate, leflunomide, cyclophosphamide, azathioprine, mertiomate, tacrolimus, cyclosporine, and biologics, including rituximab, belimumab and tetracycline;

Inclusion criteria for Systemic Sclerosis:

1. Meets 2013 ACR classification criteria for systemic sclerosis;
2. If combined with interstitial pneumonia, interstitial changes suggestive of ground-glass exudates on chest HRCT and FVC or DLCO <70% predictive value on pulmonary function tests;
3. IDefinition of relapsed and refractory disease: ineffective conventional treatment or relapse of disease activity after remission. Definition of routine treatment: use of glucocorticoids and one or more immunomodulatory drugs for more than 6 months, including antimalarials, methotrexate, leflunomide, cyclophosphamide, azathioprine, mycophenolate mofetil, tacrolimus, cyclosporine, and biologics including rituximab, belimumab, and tetanuscept;
4. Definition of progressiveness; 1) Definition of cutaneous progression: increase in mRSS >10%; 2) Definition of lung disease progression: 10% decrease in FVC or 5% decrease in FVC with 15% decrease in DLCO (OMERACT progression).

Inclusion criteria for Recurrent refractory idiopathic inflammatory myopathy:

1. Classification criteria for inflammatory myopathy in accordance with 2017 EULAR/ACR (including DM, PM, ASS, and NM);
2. For those with muscle involvement, the MMT-8 score is lower than 142 and at least two abnormalities are found in the following five core measurements (PhGA, PtGA, or extramuscular disease activity score ≥ 2 points; total HAQ score ≥ 0.25; muscle enzyme levels are 1.5 times the upper limit of the normal range);
3. Positive myositis antibodies;
4. Ineffective conventional treatment or relapse of disease activity after remission. Definition of routine treatment: Use of glucocorticoids (above 1mg/Kg/d) and cyclophosphamide, as well as any of the following immunomodulatory drugs for more than 6 months: antimalarials, methotrexate, leflunomide, cyclophosphamide, azathioprine, mertiomate, tacrolimus, cyclosporine, and biologics, including rituximab, belimumab and tetracycline.

Inclusion criteria for relapsing refractory rheumatoid arthritis:

1. Meets the diagnostic criteria of the 2010 ACR/EULAR classification. Diagnosis of moderately or severely active rheumatoid arthritis with a previous diagnosis of rheumatoid arthritis ≥ 6 months;
2. A swollen joint count of ≥ 6 (based on 66 joint counts) and a tender joint count of ≥ 6 (based on 68 joint counts) during the Screening Period;
3. C-reactive protein (CRP) ≥ 10 mg/L or erythrocyte sedimentation rate (ESR) ≥ 28 mm/h during the Screening Period;
4. EULAR definition of refractory rheumatoid arthritis:

<!-- -->

1. Failure of treatment according to EULAR recommended guidelines and failure of treatment with ≥2 b/tsDMARDs despite failure of treatment with csDMARDs. (i) unless treatment with bDMARDs/tsDMARDs is limited due to socioeconomic factors; and (ii) if treatment with csDMARDs is contraindicated, then failure of treatment with ≥2 b/tsDMARDs of different mechanisms also fulfills the condition);
2. Symptom management of RA is considered problematic by both the patient and the physician;
3. Signs suggestive of active or progressive disease if at least 1 of the following 5 items is met

   1. At least moderate disease activity (DAS28-ESR >3.2 or CDAI >10);
   2. Signs and/or symptoms suggestive of active disease;
   3. Inability to reduce glucocorticoids to less than 7.5 mg/day prednisone or equivalent;
   4. Rapid imaging progression (1-year increase of ≥5 points in van der Heijde modified Sharp score);
   5. Decreased quality of life due to RA, although RA is well controlled;
   6. Refractory rheumatoid arthritis is diagnosed if three of the above criteria are met.

Common exclusion criteria:

1. Subjects with known severe allergic reactions, hypersensitivity, contraindication to any medications during the trial (cyclophosphamide, fludarabine, tozumabs), or subjects with a history of severe allergic reactions; 2. Subjects with active or suspected fungal, bacterial, viral, or other infections that are uncontrolled or require treatment; 3. Subjects with central nervous system disorders due to autoimmune diseases or non-autoimmune diseases(including epilepsy, psychosis, organic encephalopathy syndromes, cerebrovascular accidents, encephalitis, central nervous system vasculitis); 4. Subjects with relatively serious heart diseases, such as angina pectoris, myocardial infarction, heart failure, and arrhythmia; 5. Subjects with congenital immunodeficiency diseases; 6. Subjects with malignant tumors (except for non-melanoma skin cancer and in situ cervical, bladder, and breast cancers that have been disease-free for more than 5 years); 7. Subjects with end-stage renal failure; 8. SSubjects with positive hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) and HBV DNA titer in peripheral blood higher than the upper limit of detection; subjects with positive hepatitis C virus (HCV) antibodies and positive peripheral blood HCV RNA; subjects with positive human immunodeficiency virus (HIV) antibodies; subjects with positive for syphili; 9. Subjects with mental illness and severe cognitive impairment; 10. Subjects who have received other clinical trial treatment within 3 months; 11. Pregnant or intending to conceive women; 12. In the opinion of the investigator, there are other reasons why subjects cannot be included in this study.

Exclusion criteria for relapsing refractory dry syndrome:

1. Combined cirrhosis of the liver;
2. Combination of aplastic anemia (AA), myelodysplastic syndrome (MDS), or other myeloproliferative disease (MPD).

Exclusion criteria for recurrent refractory idiopathic inflammatory myopathies:

1. Drug-induced myositis;
2. Inclusion body myositis;
3. Tumor-associated myositis (myositis occurring within 2 years of tumor diagnosis).

Exclusion criteria for relapsed refractory rheumatoid arthritis:

Functional status of rheumatoid arthritis graded at level 4 according to ACR.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-06-27 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose-Limiting Toxicity (DLT) | up to 48 weeks after infusion
  To characterize the safety of CD19 CAR NK Cells (KN5501) for Relapsed/Refractory autoimmune diseases
Incidence of Treatment Emergent Adverse Events (TEAEs) | up to 48 weeks after infusion
  To characterize the safety of CD19 CAR NK Cells (KN5501) for Relapsed/Refractory autoimmune diseases

SECONDARY OUTCOMES:
The overall response rate (ORR) | Time Frame: 1, 3, 6, 12 and 12 months after infusion
  To characterize the efficacy of CD19 CAR NK Cell (KN5501) for Relapsed/Refractory autoimmune diseases
Disease control rate (DCR) | Time Frame: 1, 3, 6, 12 and 12 months after infusion
  To characterize the efficacy of CD19 CAR NK Cell (KN5501) for Relapsed/Refractory autoimmune diseases

CONTACTS AND LOCATIONS:
Locations (1):
- Changhai Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No